CLINICAL TRIAL: NCT05727202
Title: IVD_ Starfish_Clinical Performance Study Protocol for US - Project STARFISH - PRJ0002679
Brief Title: Project STARFISH - PRJ0002679
Acronym: STARFISH
Status: Completed | Type: Observational
Sponsor: Thermo Fisher Scientific, Inc (Industry)
Collaborators: NAMSA (Other)
Responsible Party: Sponsor
Other Study IDs: PCP0127284
Record Dates: First submitted 2023-01-26; First posted 2023-02-14 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: SARS-CoV-2 Infection; Influenza A; Influenza Type B; RSV Infection
MeSH Terms: conditions — COVID-19; Respiratory Syncytial Virus Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The study population will be composed of participants suspected of a respiratory tract infection from SARS-COV-2, Influenza A/B, or RSV. For this study, 1 nasopharyngeal swab and 1 nasal swab will be collected from each participant recruited prospectively from at least three (3) collection sites located in different geographical regions in the US.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (4):
- SARS-CoV-2 infection: 50 positive samples 500 negative samples
  Interventions: Diagnostic Test: The Applied Biosystems™ TaqPath™ COVID-19, Flu A, Flu B, RSV Select Panel
- Influenza A infection: 50 positive samples 500 negative samples
  Interventions: Diagnostic Test: The Applied Biosystems™ TaqPath™ COVID-19, Flu A, Flu B, RSV Select Panel
- Influenza B infection: 30 positive samples 500 negative samples
  Interventions: Diagnostic Test: The Applied Biosystems™ TaqPath™ COVID-19, Flu A, Flu B, RSV Select Panel
- RSV infection: 30 positive samples 500 negative samples
  Interventions: Diagnostic Test: The Applied Biosystems™ TaqPath™ COVID-19, Flu A, Flu B, RSV Select Panel

INTERVENTIONS:
Diagnostic Test: The Applied Biosystems™ TaqPath™ COVID-19, Flu A, Flu B, RSV Select Panel — A multiplex real-time PCR IVD test for the qualitative detection and identification of SARS-CoV-2, influenza A virus, influenza B virus, and respiratory syncytial virus (RSV).

SUMMARY:
This is a non-interventional study to perform the clinical performance evaluation of the Starfish Test using prospectively collected matched nasopharyngeal and nasal swab samples from the same donor.

DETAILED DESCRIPTION:
The Applied Biosystems™ TaqPath™ COVID-19, Flu A, Flu B, RSV Select Panel (referred to below as "Starfish Test") aims to develop a multiplex real-time PCR IVD test for the qualitative detection and identification of SARS-CoV-2, influenza A virus, influenza B virus, and respiratory syncytial virus (RSV).

The purpose of this performance study is to evaluate the clinical performance of the Starfish Test compared with that of a comparator device using upper respiratory specimens from subjects who have provided consent to participate in the study and meet the inclusion criteria. This Clinical Performance Study Protocol (CPS Protocol) outlines the clinical sample collection and testing protocols which will be used to satisfy the FDA 510(k) study requirements in the US.

ELIGIBILITY:
Inclusion Criteria:

* Participants of all ages must meet the following inclusion criteria to be eligible for participation in the study.

  * Ability to provide informed consent or assent (as age-appropriate). Stated willingness and ability to comply with the study procedures including nasopharyngeal and anterior nasal swab collection.
  * All-comers phase: Individuals suspected to have respiratory tract infection for seven (7) or fewer days.
  * Enrichment phase: Individuals suspected to have respiratory tract infection for seven (7) or fewer days, and with a standard of care positive PCR test result within three (3) days.

Exclusion Criteria:

* Participants meeting the following criterion will be excluded from the study:

  * Suspected to have respiratory tract infection for greater than seven (7) days.
  * Patients not suspected of having a respiratory tract infection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be composed of participants suspected of respiratory tract infection from SARS-COV-2, Influenza A/B, or RSV. After a subject is determined eligible for study participation (met inclusion criteria and did not meet exclusion criteria) and has completed the institutional review board (IRB)-approved informed consent form process (or assent, as age appropriate), the subject is enrolled into the study.
Sampling Method: Probability Sample
Enrollment: 1909 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-04-02 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint | Between February 2023 and April 2024
  The primary endpoint of this clinical performance study is to meet the minimum sample positivity requirements for nasopharyngeal samples as defined by relevant regulatory guidance.

SECONDARY OUTCOMES:
Secondary Endpoint | Between February 2023 and April 2024
  The secondary endpoint of this study is to complete the clinical performance evaluation of the Starfish Test compared with that of a predicate device using Anterior nasal specimens and meet the minimum PPA and NPA requirements and acceptance criteria for each viral target as summarized in the protocol.

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Women's Health Care Research, San Diego, California
  - Medical Center for Clinical Research, San Diego, California
  - Multi-Specialty Research Associates, Lake City, Florida
  - D&H National Research Centers, Miami, Florida
  - Quantigen, Fishers, Indiana
  - KUR Research at Columbia Medical Practice, Columbia, Maryland
  - Vida Clinical Studies, Dearborn Heights, Michigan
  - MRI Global, Kansas City, Missouri
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - KUR Research at AFC Urgent Care, Hillsdale, New Jersey
  - KUR Research at AFC Urgent Care, Paramus, New Jersey
  - Mako Medical Laboratories, Henderson, North Carolina
  - Progressive Medicine of the Triad, Winston-Salem, North Carolina
  - ClinSearch, Chattanooga, Tennessee
  - Helios Clinical Research, Jackson, Tennessee
  - Helios Clinical Research, Keller, Texas
  - Granger Medical Clinic, Riverton, Utah